CLINICAL TRIAL: NCT04298736
Title: Bariatric Surgery vs. Lifestyle Modification: Effects Against Nonalcoholic Steatohepatitis Randomized Trial
Brief Title: Bariatric Surgery vs. Lifestyle Modification for NASH
Acronym: BeLEANeR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0780
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded pathologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric Surgery (Experimental): Obese patients, BMI from 30 to 45, with or without type 2 diabetes, submitted to either laparoscopic Roux-en-Y Gastric Bypass or laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: Bariatric Surgery
- Lifestyle Modification (Active Comparator): Obese patients, BMI from 30 to 45, with or without type 2 diabetes, submitted to guided diet and physical activity.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Procedure: Bariatric Surgery — laparoscopic Roux-en-Y gastric bypass or laparoscopic Sleeve Gastrectomy
  Arms: Bariatric Surgery
Behavioral: Lifestyle modification — guided low-calorie diet and physical activity.
  Arms: Lifestyle Modification

SUMMARY:
Randomized Controlled Trial comparing the effects of Bariatric Surgery vs. Lifestyle modification on NASH resolution.

DETAILED DESCRIPTION:
Patients with biopsy-proven NASH will be randomized to either bariatric surgery or lifestyle interventions. After 1-year follow-up a liver biopsy will be done to evaluate NASH resolution

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 45
* with biopsy-proven NASH
* with or without type 2 diabetes
* that fit for bariatric surgery.

Exclusion Criteria:

* borderline NASH ou cirrhosis;
* alcohol consumption (> 20 g/day for men and > 10 g/day for women, for the last 2 years);
* other hepatic diseases (such as viral hepatitis, autoimmune hepatitis, drug-induced hepatic disease, Wilson's disease, hemochromatosis);
* HIV infection;
* unable to provide informed consent;
* previous foregut or bariatric surgery;
* malignancy;
* patients that unfit for bariatric surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
NASH resolution | 12 months
  NASH resolution evaluated by liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme S Mazzini, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil